CLINICAL TRIAL: NCT00292825
Title: SCANdinavian Vasovagal SYNCope Pacemaker Investigation (SCANSYNC)
Brief Title: Effect of Closed Loop Pacemaker Treatment on Recurrent Vasovagal Syncope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Aarhus University Hospital (Other); Biotronik SE & Co. KG (Industry)
Responsible Party: Henning Mølgaard M.D., DMSc, Aarhus University Hospital, Skejby; Århus, Denmark
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: skejbyH
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2010-04-01 (Estimated); Status verified 2010-03

CONDITIONS: Vasovagal Syncope
Keywords: vasovagal syncope; syncope; cardioinhibitory syncope; neurocardiogenic syncope; pacing; closed loop pacing; tilt table
MeSH Terms: conditions — Syncope, Vasovagal; Syncope

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Device: Pacemaker treatment, pacemaker programmed as active = CLS — Pacemaker treatment with closed loop function(CLS)
Device: Pacemaker, programmed as passive = VVI 30 beats per minute (bpm) — pacemaker treatment as VVI 30 bpm

SUMMARY:
The main purpose is to prevent syncope in patients with recurrent syncopal episodes caused by malignant vasovagal faints and bradycardia. Patients are treated by a special pacemaker (closed loop stimulation [CLS]) which can potentially identify an incipient attack and prevent syncope by pacing.

DETAILED DESCRIPTION:
The treatment of patients with recurrent syncope of vasovagal origin, not precipitated by usual vasovagal factors, and not associated with structural heart disease, is unsolved. The limitations of the conducted 5 pacemaker studies are a significant placebo effect of pacemaker treatment, underpowering and lack of double blinding. The pacemaker intervention has been accelerated dual chamber pacing at the time of bradycardia, which may be too late. However, a pooling of all data indicate a beneficial effect of pacing.

Vasodilatation is an obligate element of all vasovagal syncopal episodes and in many also an early sign associated with the hyperkinetic empty left ventricle which triggers the reflex wave. The principle in closed loop stimulation (CLS) is a continuous surveillance of the impedance in the right ventricle which correlates highly with myocardial contractility. When contractility is increased significantly atrial pacing with prolonged AV delay is commenced. This principle has been used in chronotropic incompetent patients and in one small study of patients with vasovagal syncope with a positive outcome. The hypothesis is that the CLS will potentially identify an incipient vasovagal attack and be able to prevent the drop in cardiac output and bradycardia by early accelerated pacing.

Patients will be treated 12 months with active pacing (CLS) and then crossed over to 12 months with passive pacing (VVI, 30 bpm).

The study will be double blinded, only a technician will know the status of the pacemaker.

ELIGIBILITY:
Inclusion Criteria:

* A clinical problem with vasovagal syncope which motivates considerations concerning pacemaker treatment.
* A positive tilt-table test.
* Exclusion of other causes for syncope by a complete diagnostic work-up allowing only minor cardiac abnormalities
* Syncope for >= 2 years.
* Number of syncopal episodes >= 3
* At least 1 instance of syncope within the last 6 months.
* A positive tilt-table test which reproduces the clinical syncope and is associated with a clearly abnormal haemodynamic response:

  * Vasovagal Syncope International Study (VASIS) type 1 with bradycardia < 40 bpm, or
  * VASIS type 2A, or
  * VASIS type 2B
* Stable clinical condition
* Able to accept and follow the protocol and give written consent.

Exclusion Criteria:

* Conventional indication for pacemaker (i.e. atrioventricular [AV] block)
* Indication for cardiac resynchronisation therapy (i.e. left bundle branch block [LBBB])
* Documented atrial fibrillation or flutter
* Epilepsy
* Congestive heart failure
* History of myocardial infarction (MI) or angina pectoris
* Serious chronic disease, life expectancy < 3 years.
* Age < 25 years
* Pregnant and lactating women
* Participating in other investigation

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Recurrence of syncope, active (CLS pacing) versus passive (VVI=30) pacing period | 12 months + 12 months

SECONDARY OUTCOMES:
Number of syncopal and presyncopal episodes, active versus passive pacing period | 12 months+12 months
Quality of life, active versus passive pacing period | 12 months+12 months

CONTACTS AND LOCATIONS:
Overall Officials: Henning Mølgaard, MD, DMSc, Principal Investigator — Department of Cardiology, Skejby Sygehus, Aarhus University Hospital, Denmark
Locations (1):
- Henning Mølgaard, MD, DMSc, Århus N, Århus N, Denmark